CLINICAL TRIAL: NCT02767128
Title: Pharmacokinetics and Absolute Bioavailability of Fer-In-Sol (Ferrous Sulfate) and Triferic (Ferric Pyrophosphate Citrate) Administered Orally With Shohl's Solution in Healthy Volunteers
Brief Title: Pharmacokinetics and Absolute Bioavailability of Fer-In-Sol and Triferic Administered Orally With Shohl's Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMFPC-18
Record Dates: First submitted 2016-05-05; First posted 2016-05-10 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2018-08

CONDITIONS: Iron-refractory, Iron-deficiency Anemia (IRIDA)
Keywords: pharmacokinetics; healthy adult volunteer
MeSH Terms: conditions — Iron-Refractory Iron Deficiency Anemia | interventions — ferric pyrophosphate; spleen fibrinolytic proteinase (human); ferrous sulfate; Citrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Fer-In-Sol Orally (Experimental): Patients will receive A single oral dose of Fer-In-Sol at 3 mg Fe/kg body weight (bw).
  Interventions: Drug: Fer-In-Sol
- Shohl's solution followed by Fer-In-Sol Orally (Experimental): Patients will receive a single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7ml/kg bw) followed after 10 minutes by Fer-In-Sol at 3 mg Fe/kg bw.
  Interventions: Drug: Fer-In-Sol; Drug: Shohl's solution
- Triferic Orally (Experimental): Patients will receive a single oral dose of Triferic at 3 mg Fe/kg bw.
  Interventions: Drug: Triferic
- Shohl's solution followed by Triferic Orally (Experimental): Patients will receive a single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7 ml/kg bw) administered 10 minutes prior to a single oral dose of Triferic at 3 mg Fe/kg bw.
  Interventions: Drug: Triferic; Drug: Shohl's solution
- Shohl's solution followed immediately by Triferic (Experimental): Patients will receive a single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7 ml/kg bw) followed immediately by a single oral dose of Triferic at 3 mg Fe/kg bw.
  Interventions: Drug: Triferic; Drug: Shohl's solution
- Triferic via IV (Experimental): Patients will receive IV Triferic iron 6.6 mg diluted in an appropriate amount of D5W administered as a 120 mL infusion intravenously for 4 hours.
  Interventions: Drug: Triferic
- Baseline (No Intervention): baseline serum iron profile will be determined for each patient. no study drug will be administered.

INTERVENTIONS:
Drug: Triferic
  Other Names: ferric pyrophosphate citrate; FPC
  Arms: Shohl's solution followed by Triferic Orally; Shohl's solution followed immediately by Triferic; Triferic Orally; Triferic via IV
Drug: Fer-In-Sol
  Other Names: Ferrous Sulfate
  Arms: Fer-In-Sol Orally; Shohl's solution followed by Fer-In-Sol Orally
Drug: Shohl's solution
  Other Names: Oracit
  Arms: Shohl's solution followed by Fer-In-Sol Orally; Shohl's solution followed by Triferic Orally; Shohl's solution followed immediately by Triferic

SUMMARY:
The main purpose is to determine the pharmacokinetics (PK) of Triferic iron administered orally in healthy adult volunteers. It is a randomized multiple treatments, single dose study.

DETAILED DESCRIPTION:
This is a Phase 1/2, randomized multiple treatments, single dose study assessing the pharmacokinetics (PK) and absolute bioavailability of Fer-In-Sol ( Ferrous Sulfate) and Triferic (ferric pyrophosphate citrate, or FPC) administered orally with Shohl's solution in healthy volunteers.

Total participation in the study is approximately six weeks and is comprised of a screening visit, 6 treatment periods, and a follow-up visit.

The study will be conducted over a 13 day period:

Day 1 will used to determine the baseline serum iron profile for each subject.

Each subject will subsequently receive in a randomized sequence between Day 2 and 10:

1. A single oral dose of Fer-In-Sol at 3 mg Fe/kg body weight (bw).
2. A single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7 ml/kg bw) followed after 10 minutes by Fer-In-Sol at 3 mg Fe/kg bw
3. a single oral dose of Triferic PO at 3 mg Fe/kg bw
4. a single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7 ml/kg bw) administered 10 minutes prior to a single oral dose of Triferic at 3 mg Fe/kg bw.
5. a single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7 ml/kg bw) followed immediately by a single oral dose of Triferic at 3 mg Fe/kg bw.

All subjects will receive a single dose of 6.6 mg Triferic as a 4 hour IV infusion (to mimic the 4 hour iron tolerance test) on Day 12.

Blood samples will be obtained at various times to analyze for serum iron parameters and for safety.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be able to provide informed consent and have personally signed and dated the study written informed consent document before completing any study-related procedures.
2. The patient has hemoglobin, MCV and reticulocyte values within the reference range for gender. (Male: Hgb ≥13.0 g/dL; Female Hgb ≥ 12.0 g/dL) at Screening.
3. The patient must have transferrin saturation (TSAT) of ≥20% at Screening.
4. The patient must have a total iron binding capacity (TIBC) of ≥250 ug/dL at Screening.
5. The patient must have a serum ferritin within the following reference range for gender at Screening: (Males: 23-336 ng/mL; Females: 11-306 ng/mL).
6. The patient must agree to discontinue all iron preparations for 14 days prior to Baseline.
7. If the patient is female, she must be non-pregnant and non-lactating, and be at least 90 days post-partum (if applicable) at Screening. Women of childbearing potential must be willing to use appropriate birth control during the entire duration of the study.
8. The patient must be willing and able to comply with all study procedures and restrictions.
9. The patient must have no clinically significant abnormal findings on medical history, vital signs, physical examination, or clinical laboratory results during Screening.
10. The patient must have a body mass index (BMI) of ≤35.0 kg/m2 at Screening.

Exclusion Criteria:

1. The patient has had administration of oral iron supplements within 14 days prior to Baseline.
2. The patient has received IV iron within 6 months prior to Screening.
3. The patient has a serum CRP concentration above the upper limit of normal at Screening or Baseline (> 6.0 mg/L).
4. The patient has concurrent or recurrent disease (e.g., cardiovascular, renal, hepatic, gastrointestinal, malignant, etc.) that could affect the action or disposition of the investigational product utilized in this study, or could affect clinical or laboratory assessments.
5. The patient has an acute illness within 14 days prior to Baseline.
6. The patient is currently using any medication (including prescription, over-the-counter (OTC), herbal, or homeopathic preparations) within 14 days prior to Baseline. Exceptions are contraceptives, hormone replacement therapy, acetaminophen, and non-steroidal anti-inflammatory drugs.
7. The patient has known or suspected intolerance or hypersensitivity to iron-containing products.
8. The patient has a history of alcohol or substance abuse within the past year.
9. The patient has a positive screen for cotinine or drugs of abuse.
10. The patient is positive for HIV, hepatitis B, or hepatitis C by history.
11. The patient donated blood or blood products (e.g., plasma or platelets) within 30 days prior to Screening.
12. The patient has participated in an investigational drug study within 30 days prior to Screening.
13. The patient is pregnant or intends to become pregnant before completing the study.
14. The patient's current medical status, in the investigator's opinion, would preclude participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD, FACP, Study Director — Rockwell Medical, Inc
Locations (1):
- Jasper Clinic, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: This is a cross-over pharmacokinetic (PK) study where all participants underwent baseline blood sampling over 24 hours for PK purposes followed by five different oral treatments in a randomized sequence: Fer-In-Sol 3 mg Fe/kg, Shohl's solution 0.7 mL/kg followed 10 minutes later by Fer-In-Sol 3 mg Fe/kg, Triferic 3 mg Fe/kg, Shohl's solution 0.7 mL/kg followed 10 minutes later by Triferic 3 mg Fe/kg, and Shohl's solution 0.7 mL/kg followed immediately by Triferic 3 mg Fe/kg. 24 blood sampling for PK purposes took place at each randomized treatment visit. Once the randomized sequence was completed, all subjects were administered 6.6 mg Triferic intravenously at the last treatment visit, with blood sampling for PK purposes over 24 hours.
Period: Overall Study
Arm/Group | All Participants
Started | 14
Baseline | 14
Fer-In-Sol | 14
Shohl's + Fer-In-Sol | 14
Triferic | 14
Shohl's + Triferic After 10 Min | 14
Shohl's + Triferic Immediately | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: All 14 participants completed every arm of the study. Therefore, the baseline demographic characteristics of the Safety Population as a whole also reflect the characteristics of each arm of the study.
Arm/Group | Safety Population
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Body Mass Index [Mean (Standard Deviation); unit: Kilogram/square meter] | 24.5 (3.93)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of Total Iron From Triferic Administered Orally in Adult Healthy Patients: Cmax
Description: The outcome will be measured by assessing the Cmax of total iron with multiple different oral iron treatment. The following oral iron dosing treatments will be measured: Treatment A (Fer-in-Sol 3 mg iron/kg), Treatment B (Shohl's solution followed after 10 minutes by Fer-In-Sol, 3 mg/kg), Treatment C (Triferic 3 mg iron/kg), Treatment D (Shohl's solution followed after 10 minutes by Triferic 3 mg/kg), Treatment E (Shohl's solution followed immediately by Triferic 3 mg/kg), Treatment F (Triferic 6.6 mg IV over 4 hours)
Time Frame: 0, 1, 2, 4, 6, 8, 12, 16, and 24 hours
Population: 14 patients completed all six treatments. While all participants had adequate blood samples collected to be included in pharmacokinetic analysis, some samples were below the quantifiable limit (BLQ) of the bioanalytical assay, which was 50 micrograms/deciliter. Therefore, number of participants analyzed for each treatment does not equal 14.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/deciliter
Groups:
- Treatment A: Patients will receive a single oral dose of Fer-In-Sol at 3 mg Fe/kg body weight (bw).
- Treatment B: Patients will receive a single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7ml/kg bw) followed after 10 minutes by Fer-In-Sol at 3 mg Fe/kg bw.
- Treatment C: Patients will receive a single oral dose of Triferic at 3 mg Fe/kg bw.
- Treatment D: Patients will receive a single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7 ml/kg bw) administered 10 minutes prior to a single oral dose of Triferic at 3 mg Fe/kg bw.
- Treatment E: Patients will receive a single oral dose of Oracit Shohl's solution 0.67 mEq/L (0.7 ml/kg bw) followed immediately by a single oral dose of Triferic at 3 mg Fe/kg bw.
- Treatment F: Patients will receive IV Triferic iron 6.6 mg diluted in an appropriate amount of D5W administered as a 120 mL infusion intravenously for 4 hours.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 14 | 13 | 7 | 11 | 10 | 13
microgram/deciliter | 140 (39.4) | 62.0 (78.7) | 32.4 (93.9) | 51.9 (82.2) | 52.0 (71.8) | 100 (91.5)

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: The number of participants in each treatment group who experienced treatment emergent adverse events will be quantified.
Time Frame: 13 days
Population: Safety Population: all enrolled subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Participants | 7 | 5 | 2 | 6 | 6 | 2

3. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs)
Description: The number of participants in each treatment group who experienced treatment emergent serious adverse events will be quantified.
Time Frame: 13 days
Population: Safety Population: all enrolled subjects who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment F
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Fer-In-Sol Orally | Shohl's Solution Followed by Fer-In-Sol Orally | Triferic Orally | Shohl's Solution Followed by Triferic Orally | Shohl's Solution Followed Immediately by Triferic | Triferic Via IV
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 7/14 | 5/14 | 2/14 | 6/14 | 6/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fer-In-Sol Orally (N=14) | Shohl's Solution Followed by Fer-In-Sol Orally (N=14) | Triferic Orally (N=14) | Shohl's Solution Followed by Triferic Orally (N=14) | Shohl's Solution Followed Immediately by Triferic (N=14) | Triferic Via IV (N=14)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Defaecation Urgency (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Flatuence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel Puncture Site Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days